CLINICAL TRIAL: NCT03931382
Title: Evaluating Virtual Reality as an Adjunct in Procedural Preparation for Magnetic Resonance Imaging (MRI)
Brief Title: Virtual Reality Preparation for Medical Imaging
Acronym: VR-MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Children's Hospital (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, John Jacob, Executive Director & Head, Digital Lab, British Columbia Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H19-00371
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Virtual Reality; Paediatrics; Radiology

STUDY DESIGN:
Intervention Model Description: randomized, unblinded, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality (Experimental): In this arm, participants will receive 45 minutes of preparation using a simulated virtual reality experience designed in collaboration with Medical Imaging and Child Life Specialists.
  Interventions: Behavioral: Virtual Reality Simulator
- Mock MRI (Active Comparator): In this arm, participants will receive 45 minutes of preparation using the standard of care simulator, conducted by a Child Life Specialist
  Interventions: Behavioral: Mock MRI Simulator
- Manual (Active Comparator): In this arm, participants will receive 45 minutes of preparation using the standard of care MRI Preparation Booklet for non-sedated MRIs.
  Interventions: Behavioral: Standard Preparation Manual

INTERVENTIONS:
Behavioral: Virtual Reality Simulator — The VR intervention is underpinned by experiential learning and social cognitive theory, such that user will observe successful performance and simulation to encourage imitation and reinforce success in the assessment. All participants will be undergoing a simulation assessment with the head coil.
  Arms: Virtual Reality
Behavioral: Mock MRI Simulator — The mock MRI is provided by the Child Life Specialist, according to the current care plan which consists of exposing children to the MRI simulator, medical devices, and procedures. The mock MRI is located within the medical imaging facility. All participants will be undergoing a simulation assessment with the head coil.
  Other Names: Mock MRI
  Arms: Mock MRI
Behavioral: Standard Preparation Manual — The standard MRI preparation manual provides access to a series of printed photos and text showing the MRI experience step-by-step to help prepare for MRI. All participants will be undergoing a simulation assessment with the head coil.
  Arms: Manual

SUMMARY:
This pilot project aims to establish evidence to investigate whether a virtual reality intervention can be implemented to reduce anxiety and efficiently prepare children for non-sedated MRI assessments. The study consists of comparing the current modes of delivery though a mock behavioural assessment and inquiry into the acceptability and utility of the intervention components, including potential barriers to adherence or behavioural change that could have unintended consequences.

DETAILED DESCRIPTION:
Approximately 50% of pediatric patients experience elevated anxiety and distress prior to new medical procedures. This issue is critically important because it not only impacts patient experience and is associated with psychological and physiological distress, but it can affect the efficiency of medical procedures, length of hospital stay, and resource utilization - all of which have economic impacts to both families and the health system. During medical procedures specifically, anxiety can cause non-compliance or unintentional movements which often leads to failure to complete the procedure or poor image quality, necessitating multiple attempts or the use of sedation to achieve the desired quality of imaging for diagnosis.

The impact of sedating a patient has several downstream effects, including the increased potential for adverse events, as well as the need for specialized clinical staff (i.e. Anesthesiologists, Post-Anesthetic Care Nurses, etc), medications, and lengthier post-procedural monitoring. Studies have also indicated an increase in negative post-procedural clinical outcomes, such as increase pain perception, increased pharmaceutical consumption, reductions in sleep and eating, anxiety, and greater overall patient dissatisfaction.

Child Life Specialists (CLS) are specialty trained individuals that work with patients and families to improve patient experiences during stress provoking medical procedures, such as medical imaging. Procedural preparation with a CLS for MRI involves exposure to an MRI simulator. The MRI simulator appears and sounds identical to the real MRI, but lacks a magnet and thus functionality to take real images. It's suggested that this type of non-sedated preparation program can reduce anxiety and distress, ultimately reducing sedation rates.

While access to preparation programs with the CLS have improved, capacity limitations exist and there are socioeconomic costs of only having this support available on-site at BC Children's Hospital. Transportation barriers have been repeatedly identified in the literature and by parents as a source of unmet health needs for children in both rural and inner-city populations. This is significant because it a caregiver cannot get their child to the MRI simulator, they miss the opportunity for a non-sedated MRI. Consequently, resources and the risk for complications increase. As such, a virtual reality program has the capacity to increase access to patients who live afar, who are not mobile, and who need extra practice without the financial and physical limitations associated with the traditional hospital simulation.

ELIGIBILITY:
Inclusion Criteria:

* open recruitment of participants between the ages of 4-to-18 years

Please note that this trial does not include a diagnostic MRI. Participants do not need to be scheduled for a diagnostic MRI for inclusion.

Exclusion Criteria:

* mental disability
* significant visual and auditory impairment
* inability to speak or understand English
* history of seizures or epilepsy
* facial or head wounds

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Jacob, Principal Investigator — Provincial Health Services Authority British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stunden C, Stratton K, Zakani S, Jacob J. Comparing a Virtual Reality-Based Simulation App (VR-MRI) With a Standard Preparatory Manual and Child Life Program for Improving Success and Reducing Anxiety During Pediatric Medical Imaging: Randomized Clinical Trial. J Med Internet Res. 2021 Sep 22;23(9):e22942. doi: 10.2196/22942. PMID 34550072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out between July 2019 and February 2020.
Pre-assignment Details: Participants were excluded if they had mental disability, current concussion, significant visual and/or auditory impairment, inability to speak and understand English, history of seizures or epilepsy, facial or head wounds, or inability to move their head in all directions.
Groups:
- Virtual Reality: In this arm, participants will receive 45 minutes of preparation using a simulated virtual reality experience designed in collaboration with Medical Imaging and Child Life Specialists.
  Virtual Reality: The VR intervention is underpinned by experiential learning and social cognitive theory, such that user will observe successful performance and simulation to encourage imitation and reinforce success in the assessment. All participants will be undergoing a simulation assessment with the head coil.
- Mock MRI: In this arm, participants will receive 45 minutes of preparation using the standard of care simulator, conducted by a Child Life Specialist
  Simulator Preparation: The mock MRI is provided by the Child Life Specialist, according to the current care plan which consists of exposing children to the MRI simulator, medical devices, and procedures. The mock MRI is located within the medical imaging facility. All participants will be undergoing a simulation assessment with the head coil.
- Manual: In this arm, participants will receive 45 minutes of preparation using the standard of care MRI Preparation Booklet for non-sedated MRIs.
  Manual: The standard MRI preparation manual provides access to a series of printed photos and text showing the MRI experience step-by-step to help prepare for MRI. All participants will be undergoing a simulation assessment with the head coil.
Period: Overall Study
Arm/Group | Virtual Reality | Mock MRI | Manual
Started | 32 | 31 | 26
Completed | 30 | 30 | 24
Not Completed | 2 | 1 | 2
Not completed — Equipment malfunction | 2 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality | Mock MRI | Manual | Total
Number analyzed (Participants) | 30 | 30 | 24 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.27 (2.61) | 9.17 (2.65) | 8.88 (2.79) | 9.12 (2.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 11 | 33
  Male | 18 | 20 | 13 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 30 | 30 | 24 | 84
History with magnetic resonance imaging [Number; unit: participants] | 3 | 1 | 3 | 7
History with any other medical imaging [Number; unit: participants] | 13 | 15 | 12 | 43
History with magnetic resonance imaging simulator [Number; unit: participants] | 2 | 1 | 0 | 3
History with virtual reality [Number; unit: participants] | 24 | 25 | 18 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Success
Description: Movement in the MRI simulation was captured by fitting participants with a motion sensor headband (MoTrak System 1.0, Psychology Software Tools Inc). Head movement was collected at 8 samples per second, yielding approximately 3300 data points per axis per participant. The threshold for a successful MRI, as defined by the department of radiology, is approximately 3-4 mm. Consequently, if at any point during the scan the participant moved >4 mm of cumulative displacement, it was noted as a fail. Success was indicated if participants were able to complete a 6-minute head scan without surpassing 4 mm of movement at any of the 3300 data points collected. The number and percentage of participants who were successful are reported.
Time Frame: 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality | Mock MRI | Manual
Number analyzed (Participants) | 30 | 30 | 24
Participants | 9 | 14 | 12

2. Primary Outcome: Child Anxiety
Description: Child anxiety was measured with the Venham picture test (VPT; score 0-8). The level of the patient's anxiety was classified as anxiety-free (score 0), low anxiety (scores 1-3), middle anxiety (scores 4-6), and high anxiety (scores 7-8).
Time Frame: Children completed the assessment at three-time points (before preparing [T1], after preparing and upon entering the simulation room for their 6-minute scan [T2], and after the assessment [T3]).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality | Mock MRI | Manual
Number analyzed (Participants) | 30 | 30 | 24
score on a scale
  Timepoint 1 | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1]
  Timepoint 2 | 0 [0 to 1] | 1 [0 to 2] | 0 [0 to 0]
  Timepoint 3 | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 0]

3. Secondary Outcome: Caregiver/Parental Anxiety
Description: Caregiver anxiety was measured with the short State-Trait Anxiety Inventory (STAI; score 6-24), a 6-item, adapted version of the well-validated Spielberger STAI Scale. The short form of the STAI includes six statements. The range for the short STAI is 6 to 24 points, with 6 points signifying no anxiety and 24 points signifying the highest level of anxiety.
Time Frame: Parents or caregivers were asked to complete the assessment on a tablet at the same time as children (before preparing [T1], after preparing and upon entering the simulation room for their child's 6-minute scan [T2], and after the assessment [T3]).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality | Mock MRI | Manual
Number analyzed (Participants) | 30 | 30 | 24
score on a scale
  Timepoint 1 | 6.5 [6 to 10] | 7 [6 to 12] | 8 [6 to 12]
  Timepoint 2 | 6 [6 to 8] | 8 [6 to 10] | 10 [10 to 16]
  Timepoint 3 | 6 [6 to 8] | 6 [6 to 10] | 8 [6.5 to 10.5]

4. Secondary Outcome: Child Satisfaction
Description: For measuring child satisfaction, participants were asked to indicate how satisfied they were with the preparation program by pointing to a visual analog scale ranging from 0 (terrible) to 100 (fantastic).
Time Frame: Participants were asked to indicate their satisfaction after the assessment, up to 15 minutes.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality | Mock MRI | Manual
Number analyzed (Participants) | 30 | 27 | 20
score on a scale | 80 (27) | 90 (12) | 73.5 (27)

5. Other Pre Specified Outcome: Parental Usability
Description: The caregivers of our participants were prompted to provide usability feedback on the preparation materials at the end of the study. Caregivers were asked to complete the USE (Usefulness, Satisfaction, and Ease of Use) Questionnaire administered at the end of the study activities on a tablet. The USE Questionnaire is a 7-point Likert rating scale from 1-strongly disagree to 7-strongly agree. Caregivers were asked to rate the preparation program on measures related to usefulness (5-strongly disagree to 35-strongly agree), ease of use (4-strongly disagree to 28-strongly agree), ease of learning (3-strongly disagree to 21-strongly agree), and satisfaction (5-strongly disagree to 35-strongly agree).
Time Frame: Caregivers were asked to complete a questionnaire at the end of the study, after the assessment, up to 15 minutes.
Population: 1 participant in the virtual reality arm declined to do the survey; 5 participants in the mock MRI arm declined to do the survey; 4 participants in the booklet arm declined to do the survey.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Virtual Reality | Mock MRI | Manual
Number analyzed (Participants) | 29 | 25 | 20
score on a scale
  Usefulness | 31 [21 to 35] | 30 [20 to 35] | 28.5 [23 to 33]
  Easy to use | 24 [17 to 28] | 24 [16 to 28] | 24 [22 to 28]
  Easy to learn | 18 [12 to 21] | 18 [12 to 21] | 19.5 [12 to 21]
  Parental Satisfaction | 31 [23 to 35] | 31 [20 to 35] | 27 [24 to 33]

6. Other Pre Specified Outcome: Assessment Time
Description: The assessment time was defined as the time spent in the simulated MRI room until the participant was discharged from the simulation experience, either as successful or noncompliant.
Time Frame: A maximum assessment time of 20 minutes was allowed. The time spent transitioning between activities or breaks required for reasons unrelated to the study was not accounted as time.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Virtual Reality | Mock MRI | Manual
Number analyzed (Participants) | 30 | 30 | 24
Minutes | 11.79 (1.99) | 10.17 (3.44) | 11.19 (3.80)

7. Other Pre Specified Outcome: Fun
Description: Fun was measured using the Smilyometer Likert Scale, a part of the Fun Toolkit. The Smileyometer was used before and after the children interacted with a preparation program. The rationale for using it before is that it can measure their expectations and for using it afterward is that it is assumed that the child is reporting experienced fun. After allocation to a preparatory program, children were asked how good they thought the preparation would be by pointing to the Smilyometer Likert Scale to indicate their expectation of using the intervention. After using the preparation and completing the assessment (timepoint 3 [T3]), the children were again asked how good they thought the preparation actually was using the same Smileyometer Likert scale. The Smileyometer is a Likert scale from 1 (Awful) to 5 (Fantastic).
Time Frame: Participants were asked to rate expected fun at baseline and then rate the actual fun after completing the assessment [T3], up to 15 minutes.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Virtual Reality | Mock MRI | Manual
Number analyzed (Participants) | 30 | 27 | 20
score on a scale
  Expected | 4 [3 to 5] | 4 [2 to 5] | 3 [3 to 5]
  Actual | 4 [1 to 5] | 4 [1 to 5] | 4 [1 to 5]

8. Other Pre Specified Outcome: Preparation Time
Description: The preparation time started when the study staff finished describing the preparation program, and the researcher indicated that it was time to begin the active preparation. The preparation time was stopped upon indication that the participant felt ready to take the assessment. This time frame was selected as it was the allotted appointment time provided by our hospital CLP to prepare patients and their families for medical imaging procedures.
Time Frame: A maximum preparation time of 45 minutes was allowed.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Virtual Reality | Mock MRI | Manual
Number analyzed (Participants) | 30 | 30 | 24
minutes | 22.05 [20.40 to 23.69] | 15.06 [13.82 to 16.03] | 9.98 [7.76 to 12.20]

9. Other Pre Specified Outcome: Number of Participants Who Would Recommend to a Friend
Description: We asked the children if they would recommend the preparation to a friend who needed an MRI.
Time Frame: Whether the participant would recommend the preparation to a friend was asked after participants prepared for the MRI and completed the assessment [T3], up to 15 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality | Mock MRI | Manual
Number analyzed (Participants) | 30 | 27 | 20
Participants | 28 | 22 | 14

ADVERSE EVENTS:
Time Frame: Each participant was monitored while they were participating in the study components, from baseline to after the assessment [T3], up to 15 minutes. No followup occured.
Description: This was a minimum risk study.
Arm/Group | Virtual Reality | Mock MRI | Manual
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/24
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT03931382/Prot_SAP_000.pdf